CLINICAL TRIAL: NCT00856648
Title: SmartPill Monitoring for Assessment of GI Function in SCI
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: B4162C-3; KOR-09-02 (Other: James J. Peters VA Medical Center)
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: SCI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — No Biospecimens will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: SCI
  Interventions: Device: SmartPill ingestion and monitoring
- Group 2: Able-bodied
  Interventions: Device: SmartPill ingestion and monitoring

INTERVENTIONS:
Device: SmartPill ingestion and monitoring — The SmartPill device will be ingested and remotely monitored until it is excreted in a normal bowel movement.

SUMMARY:
The present study aims to evaluate the relationship between the level of SCI and the impairment of Colonic transit time (CTT) and Total transit time (TTT) by using the SmartPill device. The SmartPill, an FDA approved device, is a wireless capsule that is ingested and transmits values for GI pH, temperature, and pressure as it travels throughout the digestive system. The SmartPill can also be used to assess CTT and TTT. In comparing values for CTT, TTT, pH, temperature, and pressure in SCI patients to healthy, able-bodied controls, the SmartPill device may provide valuable insight into the pathophysiological implications of SCI on GI function. This information may allow medical professionals to provide more effective plans of care for this population, subsequentially enhancing quality and quantity of life. The SmartPill device may also provide a less invasive alternative to assessing these variables, compared to traditional modalities.

DETAILED DESCRIPTION:
Total Transit Time Total transit time (TTT) is simply the amount of time (hours) it takes for a meal to travel from the mouth, through the digestive tract and for its waste by-products to be eliminated through a bowel movement. Inter-individual TTT can vary greatly due to dietary habits, age, climate, exercise habits, immobility, medications and other lifestyle variables. Due to these multiple variables, a general TTT for the public cannot be determined. It is clear however, that a healthy person should have a total transit time ranging from 8 to 14 hours, resulting in one to three loose bowel movements every 24 hours. People who are in good physical condition, consume fiber-rich diets, and take no constipating medications are most likely to have a normal TTT. Colonic transit time (CTT) is the amount of time it takes for a partially digested meal to travel from the terminal ileum, through the large bowel and for its waste by-products to be eliminated through a bowel movement.

There are several ways to measure TTT. Each requires ingesting a tracking device or a tracer that can be monitored as it moves throughout the digestive system.

Total transit time has been traditionally measured using radiopaque markers1. This technique is simple and inexpensive and can be performed in any radiology department. Several other methods have been suggested, including the single-marker bolus technique (ingestion of markers on a specific day followed by several x-rays until all markers are passed) or multiple-marker bolus technique (ingestion of markers each day for several days followed by single or multiple abdominal x-rays). Radiopaque markers have been widely used to measure total transit. This technique provides valuable clinical information and has been proven to be reliable and reproducible.

Scintigraphy can be used as an alternative to the radiopaque marker technique for measuring TTT. The tagged material is surrounded by a substance that dissolves once it arrives at the colon. Another technique widely used in the past is the Hydrogen Breath Test which measures the transit time of the meal from the mouth to the cecum. The meal reaching the colon is indicated by a rise in the relative hydrogen content in exhaled air2,3. While many valid GI assessment techniques exist, many are invasive and impose many inconveniences for patients.

A relatively new device, the SmartPill, offers the ability to assess many GI variables including temperature, pressure, pH, and transit time while minimizing the invasive nature of investigation. The SmartPill is a small wireless capsule that is ingested by the patient. Values for pressure, temperature, and pH are transmitted continuously from the capsule to a receiver carried by the patient until the capsule is excreted during normal evacuation. This information is then downloaded onto a master computer and expressed graphically for comparative purposes.

Purpose of measuring TTT Measuring TTT is useful in evaluating patients with constipation, abdominal bloating, and refractory irritable bowel syndrome. It provides quantitative information about total transit, enables the identification and characterization of transit abnormalities, and allows assessment of the severity of the problem as well as the response to therapy.

Disorders Affecting TTT Intestinal Motility Disorder (IMD) may be due to primary or secondary causes depending on endogenous or exogenous etiologies. This would include several asymptomatic conditions, such as maldigestion, achalasia, or alkaline bile reflux from the duodenum to the stomach. Intestinal pseudo-obstruction (Ogilvie syndrome), irritable bowel syndrome (IBS), fecal incontinence, and constipation are all conditions related to disordered intestinal motility. Many common drugs (tricyclic antidepressants, diuretics, laxatives, lithium salts, vinca alkaloids, chemotherapy agents, etc.) may interfere with intestinal motility on the receptor level or by interfering with the parasympathetic nervous system, which largely controls GI motility. Drugs such as benzodiazepines, lithium salts, laxatives, and codeine cause secondary stasis4. The latter can produce narcotic bowel syndrome, which is usually observed in patients who abuse opiates for chronic pain. Endocrine disorders, such as myxedema, can also cause gastrointestinal obstruction due to the decrease in the thyroid hormone level as well as an imbalance in sodium and potassium metabolism.

CTT in SCI patients The magnitude of bowel dysfunction in spinal cord injury patients has been documented in several studies. Spinal cord injury affects colorectal motility, transit times, and bowel emptying, often leading to constipation, fecal incontinence or a combination of the two. Although these symptoms are not life-threatening, they may negatively impact quality of life as well as increase levels of anxiety and depression5.

Abnormal bowel function is one of the most bothersome problems in patients with SCI. While it is known how bowel dysfunction affects quality of life, research examining the pathophysiological causes of bowel dysfunction are limited. Moreover, most studies have provided only partial information on bowel dysmotility, focusing on only CTT or anal dysfunction, rather than identifying a comprehensive neurogenic bowel pattern according to different neurological abnormalities and clinical manifestations.

Constipation, obstructive defecation, and fecal incontinence are known to be frequent complications in SCI. However, their presence and severity are not homogeneous in all patients and depend on the integration of mechanisms such as abdominal compression, colorectal motor activity, and anal sphincter function as well as digitalization for bowel evacuation. Paralleling these complications, CTT is increased in SCI subjects when compared with the normal populations. Recent clinical studies of individuals with SCI have identified prolonged CTT in 57% of the subjects6. While these studies investigated the correlation between intestinal symptoms and the level of SCI, the relationship between intestinal symptoms and the changes in CTT were not evaluated. While several studies have identified prolonged CTT in SCI patients, other investigations have not produced consistent findings7, 8.

The present study aims to evaluate multiple variables of GI function in both patients with SCI and able-bodied controls using the SmartPill device. In comparing values for TTT, CTT, pH, temperature, and pressure in patients with SCI to healthy, able-bodied controls, the SmartPill device may provide valuable insight into the pathophysiological implications of SCI on GI function.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 75
* Spinal cord lesion at any level at least 6 months from injury
* The patient is able to understand the treatment and is willing to comply with the prescribed regimen
* At least one or more of the following symptoms:
* Bowel program >30 minutes
* Episodes of fecal incontinence once or more per month

Exclusion Criteria:

* Inadequately managed complications related to SCI
* Evidence of bowel obstruction
* Evidence of inflammatory bowel disease
* History of cerebral palsy or cerebral apoplexy
* Multiple sclerosis
* Diabetic polyneuropathy
* Previous abdominal or perianal surgery including Hernia repair , total polyp removal (not including minor surgery as appendectomy or haemorrhoidectomy)
* Pregnant or lactating
* Evidence of spinal shock
* Mentally unstable
* Treatment with more than 5 mg prednisolon per day.
* PNS implant (sacral nerve stimulation)
* History of gastric ulcers
* Disorders of swallowing
* Suspected strictures, fistulas or physiological GI obstruction.
* GI surgery within past three months
* Severe dysphagia to food or pills
* Crohns disease or diverticulitis
* Use of implanted or portable electro-mechanical medical devices such as cardiac pacemakers or infusion pumps.
* Known intolerance to the SmartPill device
* Known food allergies to any component of the standard meal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SCI and able-bodied individuals, 18-75 years of age
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Colonic transit time (CTT) | 1-4 days

SECONDARY OUTCOMES:
Total transit time (TTT) | 1-4 days
Gastric emptying time (GET) | 1-10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Korsten, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States